CLINICAL TRIAL: NCT00990925
Title: Lifestyle Modification for Weight Loss in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cenk Tek, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0903004806; R01MH080048 (NIH)
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Schizophrenia; Schizoaffective Disorder
Keywords: Obesity; Schizophrenia; Schizoaffective disorder; weight loss
MeSH Terms: conditions — Obesity; Schizophrenia; Psychotic Disorders; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight Loss Education Group (Experimental): Involvement in weekly manualized, educational group on nutrition and lifestyle modifications to help with weight loss.
  Interventions: Behavioral: Nutritional Lifestyle Modification Group
- Usual Care (Other): Treatment as usual
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Nutritional Lifestyle Modification Group — Manualized group treatment to educate about basic nutritional concepts to help improve eating choices with the goal of losing weight.
  Arms: Weight Loss Education Group
Other: Usual Care — Care as usual
  Arms: Usual Care

SUMMARY:
The purpose of this study is to find out how effective lifestyle modification group therapy is on reducing body weight when compared to usual care in individuals with schizophrenia and/or schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be between 18 and 65 years of age.
2. Have a BMI of 28 or greater.
3. Meet DSM-IV criteria for schizophrenia or schizoaffective disorder.
4. Be on a stable dose of antipsychotic medication for at least one month, with positive symptoms stability as judged by the clinical team and investigator.

Exclusion Criteria:

1. A history of dementia or mental retardation.
2. Not capable of giving informed consent for participation in this study.
3. Ongoing pregnancy.
4. Living in a structured environment where the meals are provided as part of the program, e.g., a group home, nursing home, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is change in body weight from baseline. | 16 weeks, 6 month follow-up

SECONDARY OUTCOMES:
Change in lab values from baseline (fasting serum glucose, glycosylated hemoglobin, insulin, LDL cholesterol, triglyceride levels) | 16 weeks, 6 month follow-up
Change in questionnaires and assessments (Q-LES-Q, QLS, PANSS, Food craving scales, Food frequency scales, Food preference scales) | 16 weeks, 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States